CLINICAL TRIAL: NCT05483777
Title: Investigation of the Effect of Platelet Rich Fibrin (PRF) Application on Wound Healing in Diabetic Foot Wound
Brief Title: Application of Platelet-Rich Fibrin on Diabetic Foot Wound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ebru ÇELEBİ, Lecturer, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AIBU-HEM-EC-01
Record Dates: First submitted 2022-07-28; First posted 2022-08-02 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Foot
Keywords: Diabetic Foot; Platelet-Rich Fibrin; Wound Healing
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: It is planned to include 7 patients for the experimental group and 7 patients for the control group (14 patients in total) in this research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF (Experimental): If the patient is in the experimental group, platelet rich fibrin will be applied to the diabetic foot wound.
  Interventions: Procedure: PRF
- CWD (No Intervention): If the patient is in the control group, classic wound dressing will be applied to the diabetic foot wound.

INTERVENTIONS:
Procedure: PRF — Platelet-rich fibrin preparation and application technique will applied to the experimental group.
  Arms: PRF

SUMMARY:
This study was planned as a prospective case-control study to examine the effect of PRF application on wound healing in diabetic foot wound. The sample of the study will consist of patients with diabetic foot wounds, who met the inclusion criteria and agreed to participate in the study. It is planned to include 7 patients for the experimental group and 7 patients for the control group (14 patients in total). If the patient is in the experimental group, PRF will be applied to the diabetic foot wound, and in the control group, classic wound dressing (CWD) will be applied.

DETAILED DESCRIPTION:
Foot ulcer is a common complication in diabetic patients, in some cases requiring hospitalization and may result in amputation. Effective treatment and care of diabetic foot is as important as prevention. For this reason, the condition of the wound should be evaluated well, effective wound care materials should be used, and current evidence-based practices should be included in treatment and care. One of these current applications is PRF. In the literature, the success and positive effects of PRF applications on dentistry, plastic surgery, orthopedics, eye surgery, diabetic foot, chronic arterial and venous ulcers, and complex wounds that are difficult to heal have been reported.

This study was planned as a prospective case-control study to examine the effect of PRF application on wound healing in diabetic foot wound. The population of the study will consist of patients with diabetic foot wounds, who applied to Bolu Home Health Services affiliated to the Republic of Turkey Ministry of Health Bolu Provincial Health Directorate, and who were followed up in the center of Bolu.

The sample of the study will consist of patients with diabetic foot wounds, who met the inclusion criteria and agreed to participate in the study. It is planned to include 7 patients for the experimental group and 7 patients for the control group (14 patients in total). Before starting the study, patients will be randomized in a computer program (random.org). According to the randomization results of the program, the patients in the first column will be the experimental group and the patients in the second column will be the control group. If the patient is in the experimental group, PRF will be applied to the diabetic foot wound, and in the control group, classic wound dressing (CWD) will be applied.

PRF Preparation and Application Technique (To be applied to the experimental group):

10 ml blood will be collected into a tube without anticoagulant with an injector or a vacutainer directly, from the patients included in the experimental group. Then, centrifugation will be carried out immediately at 3000 (rpm) speed for 10 minutes. This process will be applied by the researcher next to the patient by using a Yuda 800D brand desktop type centrifuge device with 6 tube capacity, 500-4000 rpm speed setting and 5-30 minutes time setting. After this procedure, the tube will be removed from the device and the PRF clot formed in the middle of the tube will be removed with forceps. This clot will be compressed into a membrane between two sterile gauzes moistened with saline, with as little finger pressure as possible. The shaped PRF will be placed to cover the entire diabetic foot wound under sterile conditions. Then the dressing will be closed by covering with sterile gauze.These applications will be repeated weekly and applied for a total of 11 weeks.

Classic Wound Dressing Application:

Classic dressing will be applied to the diabetic foot wound of the patients in the control group by the researcher. After the diabetic foot wound is evaluated, it will be irrigate with saline on sterile conditions, cover with sterile gauze and fix with a plaster. This dressing will be repeated weekly and applied for a total of 11 weeks.

Wound evaluation will be done at 1st (first day of application), 2nd, 4th, 8th and 12th weeks. "Data collection form", "Wound observation and evaluation form", 'Diabetes Self-Efficacy Scale', 'Diabetic Foot Care Self-Efficacy Scale', 'Medical Adherence Report Scale' will be used in the data collection phase of the research. The evaluation of both feet in terms of diabetic foot will be made using the 'Diabetic Foot Evaluation Form'. In addition, diabetic foot care training will be given to all patients at the first meeting.

In the power analysis (G*Power 3.1.9.4) made considering the studies in the literature, it was determined that at least 12 patients (6 experiment, 6 control) should be reached for the study. Problems that may arise with the participants during the study were taken into account, and it is planned to include at least 7 patients (14 in total) for each group, by overestimating 1 person for each of the two groups. The data will be evaluated using a statistical package program. Evaluation will be made by using various tests (dependent/independent t-test, Mann Whitney U, Wilcoxon, Kruskal Wallis, Dependent/Independent ANOVA, Friedman, etc.) and correlation tests, depending on whether the data show a normal distribution with descriptive statistical methods. The significance level to be used was determined as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* 1st or 2nd degree diabetic foot wound according to Wagner classification
* Absence of infection in diabetic foot wound
* Being over 18 years old
* Willingness to participate in the research
* Absence of any allergic disease
* Absence of bleeding disorder
* Not receiving corticosteroid treatment
* Not using anticoagulant medication
* Not smoking
* Absence of circulatory disorders in the lower extremities
* HbA1c value below 12% (Mean blood glucose value 298 mg/dL) in the most recent examination

Exclusion Criteria:

* 3rd, 4th and 5th degree diabetic foot wound according to Wagner classification
* Presence of infection in diabetic foot wound
* Being under the age of 18
* Not being willing to participate in the research
* Presence of any allergic disease
* Having a bleeding disorder
* Being on corticosteroid treatment
* Using anticoagulant medication
* Smoking
* HbA1c value above 12% (average blood glucose value 298 mg/dL) in the most recent examination
* Having circulatory disorders in the lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Wound Observation and Evaluation Form | Healing on diabetic foot wounds at 12 weeks.
  The length, width, depth, exudate, necrotic tissue, wound bed, skin around the wound, etc. aspects will be evaluated with this form.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu İLÇE, Ph.D, Study Director — Abant Izzet Baysal University; Muhammed Emin DEMİRKOL, M.D., Study Director — Abant Izzet Baysal University; Ebru ÇELEBİ, MSc, Principal Investigator — Abant Izzet Baysal University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lorig K, Ritter PL, Villa FJ, Armas J. Community-based peer-led diabetes self-management: a randomized trial. Diabetes Educ. 2009 Jul-Aug;35(4):641-51. doi: 10.1177/0145721709335006. Epub 2009 Apr 30. PMID 19407333
- [Background] Mankan T, Erci B, Bahcecioglu Turan G, Akturk U. Turkish validity and reliability of the Diabetes Self-Efficacy Scale. Int J Nurs Sci. 2017 May 4;4(3):239-243. doi: 10.1016/j.ijnss.2017.05.001. eCollection 2017 Jul 10. PMID 31406747
- [Background] Quarles BE. Educational methods increasing self-efficacy for the management of foot care in adults with diabetes and implementation of foot care behaviors, (Dissertation), Doctor of Philosophy in The College of Education at The University of Kentucky, Lexington, Kentucky; 2005
- [Background] Kır Biçer E. Enç N. Diyabetik Ayak Bakımı Özetkililik Ölçeğinin geçerlik ve güvenirlik çalışması. Diyabet, Obezite ve Hipertansiyonda Hemşirelik Forumu. 2014;6(2):40-5.
- [Background] Horne R, Hankins M. The Medication Adherence report Scale (MARS), 2001. (manuscript submitted for publication).
- [Background] Şen, E. T., Berk, Ö. S., & Sindel, D. (2019). İlaç Uyumunu Bildirim Ölçeği'nin Türkçe Uyarlamasının Geçerlik ve Güvenirlik Çalışması. İstanbul Tıp Fakültesi Dergisi, 82(1), 52-61.
- [Background] Pinto NR, Ubilla M, Zamora Y, Del Rio V, Dohan Ehrenfest DM, Quirynen M. Leucocyte- and platelet-rich fibrin (L-PRF) as a regenerative medicine strategy for the treatment of refractory leg ulcers: a prospective cohort study. Platelets. 2018 Jul;29(5):468-475. doi: 10.1080/09537104.2017.1327654. Epub 2017 Jul 20. PMID 28727481
- [Background] Somani A, Rai R. Comparison of Efficacy of Autologous Platelet-rich Fibrin versus Saline Dressing in Chronic Venous Leg Ulcers: A Randomised Controlled Trial. J Cutan Aesthet Surg. 2017 Jan-Mar;10(1):8-12. doi: 10.4103/JCAS.JCAS_137_16. PMID 28529414
- [Background] Ozer K, Colak O. Leucocyte- and platelet-rich fibrin as a rescue therapy for small-to-medium-sized complex wounds of the lower extremities. Burns Trauma. 2019 May 6;7:11. doi: 10.1186/s41038-019-0149-0. eCollection 2019. PMID 31080838
- [Background] Londahl M, Tarnow L, Karlsmark T, Lundquist R, Nielsen AM, Michelsen M, Nilsson A, Zakrzewski M, Jorgensen B. Use of an autologous leucocyte and platelet-rich fibrin patch on hard-to-heal DFUs: a pilot study. J Wound Care. 2015 Apr;24(4):172-4, 176-8. doi: 10.12968/jowc.2015.24.4.172. PMID 25853474
- [Background] Yuvasri G, Rai R. Comparison of Efficacy of Autologous Platelet-Rich Fibrin versus Unna's Paste Dressing in Chronic Venous Leg Ulcers: A Comparative Study. Indian Dermatol Online J. 2020 Jan 13;11(1):58-61. doi: 10.4103/idoj.IDOJ_119_19. eCollection 2020 Jan-Feb. PMID 32055510
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part I: technological concepts and evolution. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e37-44. doi: 10.1016/j.tripleo.2005.07.008. Epub 2006 Jan 19. PMID 16504849